CLINICAL TRIAL: NCT04855656
Title: Phase 1/1b Study of the Safety, Pharmacokinetics, Pharmacodynamics and Preliminary Clinical Activity of Lunresertib Alone or in Combination With RP-3500 or Debio 0123 in Patients With Advanced Solid Tumors
Brief Title: Study of Lunresertib Alone or in Combination With RP-3500 or Debio 0123 in Patients With Advanced Solid Tumors
Acronym: MYTHIC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Debio 0123-106; RP-6306-01 (Other: Repare Therapeutics)
Record Dates: First submitted 2021-04-09; First posted 2021-04-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1: Lunresertib Single-Agent, Dose Escalation and Food-effect Study (Experimental): Patients receive lunresertib orally until disease progression, unacceptable toxicity, or investigator/patient decision. Dose escalation will proceed until a maximum tolerated dose is identified.
  Interventions: Drug: Lunresertib
- Phase 1: Lunresertib in combination with RP-3500, Dose Escalation Study (Experimental): Patients receive lunresertib with RP-3500 orally until disease progression, unacceptable toxicity, or investigator/patient decision. Dose escalation will proceed until a maximum tolerated dose is identified.
  Interventions: Drug: Lunresertib; Drug: RP-3500
- Phase 1: Lunresertib in combination with Debio 0123, Dose Escalation Study (Experimental): Patients receive lunresertib with Debio 0123 orally until disease progression, unacceptable toxicity, or investigator/patient decision. Dose escalation will proceed until a maximum tolerated dose is identified.
  Interventions: Drug: Lunresertib; Drug: Debio0123

INTERVENTIONS:
Drug: Lunresertib — Oral PKMYT1 Inhibitor
Drug: RP-3500 — Oral ATR Inhibitor
  Arms: Phase 1: Lunresertib in combination with RP-3500, Dose Escalation Study
Drug: Debio0123 — Oral WEE1 Inhibitor
  Arms: Phase 1: Lunresertib in combination with Debio 0123, Dose Escalation Study

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of lunresertib alone and in combination with RP-3500 or in combination with Debio 0123 in patients with eligible advanced solid tumors, determine the maximum tolerated dose (MTD) and assess preliminary anti-tumor activity.

DETAILED DESCRIPTION:
Phase 1/1b, multi-center, open-label, dose-escalation study to:

* Evaluate the safety profile and MTD of lunresertib alone and in combination with RP-3500 or in combination with Debio 0123 when administered orally to establish the recommended Phase 2 dose and schedule
* Characterize the PK and pharmacodynamics of lunresertib alone and in combination with RP-3500 or in combination with Debio 0123
* Assess preliminary anti-tumor activity associated with lunresertib alone and in combination with RP-3500 or in combination with Debio 0123

This study was previously posted by Repare Therapeutics. In September 2025, sponsorship of the trial was transferred to Debiopharm International S.A

ELIGIBILITY:
Inclusion Criteria:

* Male or female and ≥12 years-of-age at the time of informed consent.
* Lansky performance status ≥50% for patients ≤16 years of age, or ECOG score of 0, 1, (or 2 for module 1) for patients >16 years of age.
* Locally advanced or metastatic resistant or refractory solid tumors.
* Patients <18 years of age must weigh at least 40 kg.
* Submission of available tumor tissue at screening or willingness to have a biopsy performed if safe and feasible
* Next generation sequencing (NGS) report obtained in a CLIA-certified or equivalent laboratory demonstrating eligible tumor biomarker.
* CCNE1 amplification (non-equivocal) as determined by either a tumor or plasma NGS test, or FISH
* FBXW7 deleterious mutations identified by either a tumor or plasma NGS test
* PPP2R1A deleterious mutations identified by either a tumor or plasma NGS test
* Measurable disease as per RECIST v1.1. For certain modules, patients with prostate cancer or ovarian cancer that have non-measurable disease but have elevated tumor markers (PSA or CA-125, respectively) can also be eligible
* Ability to swallow and retain oral medications.
* Acceptable hematologic and organ function at screening.
* Negative pregnancy test (serum) for women of childbearing potential (WOCBP) at Screening.
* Resolution of all toxicities of prior therapy or surgical procedures.
* Any prior radiation must have been completed at least 7 days prior to the start of study drugs, and patients must have recovered from any acute adverse effects prior to the start of study treatment.

Exclusion Criteria:

* Chemotherapy or small molecule antineoplastic agent given within 21 days or <5 half-lives, whichever is shorter, prior to first dose of study drug.
* History or current condition, therapy, or laboratory abnormality that might confound the study results or interfere with the patient's participation for the full duration of the study treatment.
* Patients who are pregnant or breastfeeding.
* Life-threatening illness, medical condition, active uncontrolled infection, or organ system dysfunction or other reasons which, in the investigator's opinion, could compromise the participating patient's safety.
* Major surgery within 4 weeks prior to first dose of lunresertib.
* Uncontrolled, symptomatic brain metastases.
* Uncontrolled hypertension.
* Certain prior anti-cancer therapy
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol and/or follow-up procedures outlined in the protocol.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 464 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of lunresertib either in monotherapy or in combination with RP-3500 or with Debio 0123 in patients with eligible advanced solid tumors | Up to 90 days after last administration of study intervention
  Assessed by treatment-emergent adverse events (TEAEs), physical examinations (PEs), safety laboratory assessments, electrocardiograms (ECGs), and vital sign measurements
To define the MTD of lunresertib monotherapy, and determine a recommended Phase 2 dose (RP2D) and preferred schedule | Up to 90 days after last administration of study intervention
  Assessed by the incidence of Dose-limiting toxicities (DLTs) and the incidence and severity of cumulative safety data
To define the MTD of lunresertib in combination with RP-3500 or in combination with Debio 0123, and determine a recommended Phase 2 dose (RP2D) and preferred schedule | Up to 90 days after last administration of study intervention
  Assessed by the incidence of dose-limiting toxicities (DLTs) and the incidence and severity of cumulative safety data
The relative bioavailability of lunresertib capsule formulation as compared to lunresertib tablet formulation in the fasted state | Time 0 (time of dosing) to 72 hours post-dose for each treatment condition
  Assessed by the plasma concentrations of lunresertib with calculation of pharmacokinetic (PK) parameters including maximum observed plasma concentration (Cmax), time to maximum observed plasma concentration (Tmax), area under the plasma concentration-time curve (AUC) , for both formulations in the fasted state.
The effect of food on the PK of tablet formulation of lunresertib when administered in fed conditions compared to administration under fasted conditions | Time 0 (time of dosing) to 72 hours post-dose for each treatment condition
  Assessed by the plasma concentrations of lunresertib with calculation of the ratio of PK parameters (e.g., Cmax and AUC) between the tablet formulation under fasted and fed state.
To assess the safety and tolerability of lunresertib tablets in combination with RP-3500, confirm the MTD of lunresertib tablets in combination with RP-3500, and determine a RP2D and preferred schedule | Up to 90 days after last administration of study intervention
  Assessed by DLTs, TEAEs, safety laboratory assessments, the incidence of DLTs and the incidence and severity of cumulative safety data

SECONDARY OUTCOMES:
The plasma concentrations of lunresertib monotherapy (capsule formulation) in the fasted and fed states | Up to 90 days after last administration of study intervention
  Assessed by the plasma concentrations of lunresertib with calculation of maximum observed plasma concentration (Cmax), time to maximum observed plasma concentration (Tmax), minimum observed plasma concentration (Cmin), area under the plasma concentration-time curve (AUC), elimination half-life (t1/2), and other parameters as appropriate
To assess the relationship between pharmacodynamic biomarkers and PK of lunresertib at different dose levels and/or schedules | Up to 90 days after last administration of study intervention
  Assessed by evaluation of biomarkers in pre- and on-treatment biopsies, and circulating tumor DNA (ctDNA) dynamics during treatment
The plasma concentrations of lunresertib and RP-3500 when dosed in combination | Up to 90 days after last administration of study intervention
  Assessed by the plasma concentrations of lunresertib and RP-3500 with calculation of maximum observed plasma concentration (Cmax), time to maximum observed plasma concentration (Tmax), minimum observed plasma concentration (Cmin), area under the plasma concentration-time curve (AUC), elimination half-life (t1/2), and other parameters as appropriate for each analyte
To assess preliminary anti-tumor activity achieved with lunresertib monotherapy, lunresertib in combination with RP-3500 or lunresertib in combination with Debio 0123 | Through Study Completion, an average of 1 year
  Measured by best percent change in tumor size from baseline, objective response rate (ORR), overall response rate, tumor marker response, duration of response (DOR), clinical benefit rate (CBR), progression-free survival (PFS).
To assess the safety and anti-tumor effects of lunresertib capsule + RP-3500 | Through Study Completion, an average of 1 year
  As measure by TEAEs, safety laboratory assessments, Best percent change in tumor size from baseline, ORR, overall response rate, DOR, CBR, tumor marker response, PFS
To further characterize the PK of lunresertib tablets and assess preliminary anti-tumor | Through Study Completion, an average of 1 year
  Measured by Plasma concentrations of lunresertib with calculation of Cmax, Tmax, AUC, elimination t1/2, and other PK parameters as appropriate, Best percent change in tumor size from baseline, ORR, overall response rate, DOR, CBR, tumor marker response, PFS

CONTACTS AND LOCATIONS:
Locations (22):
- United States (17):
  - #1016, Mayo Clinic, Phoenix, Arizona
  - # 1019, UCLA, Westwood Cancer Center, Los Angeles, California
  - #1025, University of California San Francisco, San Francisco, California
  - #1012, Yale, New Haven, Connecticut
  - #1017, Mayo Clinic, Jacksonville, Florida
  - #1002, Dana Farber Cancer Institute, Boston, Massachusetts
  - #1023, START Midwest, Grand Rapids, Michigan
  - #1011, Washington University, St Louis, Missouri
  - #1032, Northwell Health Cancer Institute, New Hyde Park, New York
  - #1008, Columbia University, New York, New York
  - #1004, Memorial Sloan Kettering Cancer Institute, New York, New York
  - #1010, University of Pennsylvania, Philadelphia, Pennsylvania
  - #1007, Rhode Island Hospital, Providence, Rhode Island
  - #1030, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - #1001, The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - #1013, The University of Utah, Salt Lake City, Utah
  - #1027, University of Virginia, Charlottesville, Virginia
- Canada (3):
  - #2002, The Hospital for Sick Children, Toronto, Ontario
  - #2001, Princess Margaret Cancer Centre, Toronto, Ontario
  - #2003, The Research Institute of the McGill University Health Centre, Montreal, Quebec
- #4001, Rigshospitalet - Blegdamsvej, Copenhagen, Denmark
- #3003, Sarah Cannon Research Institute, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No